CLINICAL TRIAL: NCT06836479
Title: Validation of NOURISH Project's Culturally Tailored Meals on Postprandial Glycemic Response Using Continuous Glucose Monitoring: A Quantitative and Qualitative Study
Brief Title: Using Continuous Glucose Monitoring to Quantify the Effects of NOURISH's Culturally Modified Meals on Asian Americans With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Tastermonial Inc (Industry)
Responsible Party: Principal Investigator, Minal Moharir, Clinical Assistant Professor, Medicine - Primary Care and Population Health, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 78525
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Type 2 Diabetes
Keywords: Type 2 Diabetes; Asian American; Asian Indian; Filipino; Medically Tailored Meals; Culture; Culturally Tailored Meals; Continuous Glucose Monitoring; Nutritional Interventions; Dietary Adherence; Diabetes Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Selected Diet to NOURISH Diet (Experimental): Participants in this arm will be consuming self-selected meals (baseline/control) first (During Week 2 of the intervention), followed by the NOURISH diet in the next week (Week 3). Participants will be required to fill out a food diary and questionnaires using the Tastermonital app.
  Interventions: Other: NOURISH Diet; Other: Self-Selected Diet (Control)
- NOURISH Diet to Self-Selected Diet (Experimental): Participants in this arm will be consuming the NOURISH diet first (During Week 2 of the intervention), followed by their self-selected diet (baseline/control) in the next week (Week 3). Participants will be required to fill out a food diary and questionnaires using the Tastermonital app.
  Interventions: Other: NOURISH Diet; Other: Self-Selected Diet (Control)

INTERVENTIONS:
Other: NOURISH Diet — NOURISH meals will be prepared by NOURISH chefs for seven days. Both South Asian and Filipino meal plans will be prepared, vegetarian, vegan and non-vegetarian options available for all. Participants will pick-up NOURISH meals at a Stanford facility and consume three meals (breakfast, lunch, and dinner) and two snacks over one week. There will be no caloric restriction, the calories in each meal will be informed by the average intake for the participants gender and BMI.
  Other Names: NOURISH-modified meals; NOURISH meals
Other: Self-Selected Diet (Control) — The participants will eat their routine meals without any involvement of the investigators. Participants will be required to wear the CGM during this time and keep a detailed food log through Tastermonial.
  Other Names: Routine Diet; Baseline; Control

SUMMARY:
The investigators are hoping to determine whether tailoring the diet of someone with type 2 diabetes to their ethnic group while following American Diabetes Association guidelines can make a significant difference in their blood sugar controls. Participants will be required to wear a Continuous Glucose Monitor (CGM) for 1-month so that the investigators can compare blood sugar levels when participants are eating their routine diet vs. the culturally tailored diabetes diet.

DETAILED DESCRIPTION:
This clinical trial evaluates the impact of culturally tailored, American Diabetes Association (ADA)-compliant meals on the glycemic control of Asian Indian and Filipino individuals with Type 2 Diabetes Mellitus (T2DM). This study leverages a crossover design to compare glycemic responses during two distinct dietary phases: a self-selected diet phase (baseline/control/routine diet) and an intervention phase featuring NOURISH meals. NOURISH Meals will be delivered to designated pick-up points on the Stanford campus and Stanford clinics. Participants will be equipped with Continuous Glucose Monitors (CGMs) to track glucose trends across the study and will be required to keep a food log through Tastermonial, enabling detailed analysis of postprandial glucose responses and key metrics.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as Asian Indian or Filipino
* Diagnosed with T2DM
* Can pick up meals from a designated area on the Stanford Campus
* Willing to wear a CGM for 30 days

Exclusion Criteria:

* Currently taking insulin, GLP -1 and SGLT 2
* Known severe allergic reactions and/or food intolerances that would interfere with the ability to eat
* Those who, in the opinion of the investigators, cannot reliably complete the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Positive Area Under the Curve (pAUC) for Blood Glucose | During Week 2, Week 3
  Upon analysis of the CGM data graphs, the area under the curve will be analyzed. The goal is to observe the difference in glucose levels when participants consume NOURISH meals versus the self-selected diet. Higher pAUC values indicate higher average blood glucose and possibly decreased glycemic control, whereas lower pAUC values indicate lower average blood glucose and possibly increased glycemic control.

SECONDARY OUTCOMES:
Glucose % Time in Range Over the Course of the Intervention as Compared to the Baseline | During Week 2, Week 3, Week 4
  Using the glucose readings from the continuous glucose monitors, the daily glucose values for participants will be plotted. Analysis will be done to identify the %-proportion of time participant's glucose levels fall within a pre-specified range. Area values for both the self-selected diet and NOURISH diet will be compared for each participant and tested for statistical significance. Higher glucose %-time in range indicates that the glucose fell within a certain range for a larger portion of time, lower glucose %-time in range indicates that glucose deviated out of the specified range.
Adherence to NOURISH Diet | 1 week
  Participants will be performing journal logs throughout the study via the Tastermonial app. They will be required to upload information on how much of the meal they consumed and if they replaced the NOURISH meal with a self-selected one for any reason. Analysis will be conducted to understand the number of meals and days participants adhered to NOURISH meals and the blood glucose levels measured.
  Question asked to participants: "What proportion of this meal did you consume?"
  Answer choices: "I did not eat this meal at all", "25%", "50%". "75%", "I finished the full meal"

CONTACTS AND LOCATIONS:
Overall Officials: Minal Moharir, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No